CLINICAL TRIAL: NCT01717703
Title: Effect of Sugars-Sweetened Commercial Beverages on Short-Term Food Intake Regulation in Normal Weight and Overweight/Obese 9-14 Year Old Boys and Girls
Brief Title: Sugars-sweetened Commercial Beverages on Short-term Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Assisstant Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2009-020-001
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
Keywords: prevention
MeSH Terms: conditions — Obesity | interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Water Control (Experimental): Water Control
  Interventions: Dietary Supplement: Water
- Fruit drink (Experimental): Fruit drink
  Interventions: Dietary Supplement: Fruit drink
- Cola (Experimental): Cola
  Interventions: Dietary Supplement: Cola
- 1% chocolate milk (Experimental): 1% chocolate milk
  Interventions: Dietary Supplement: 1% chocolate milk

INTERVENTIONS:
Dietary Supplement: Water
  Arms: Water Control
Dietary Supplement: Fruit drink
  Arms: Fruit drink
Dietary Supplement: Cola
  Arms: Cola
Dietary Supplement: 1% chocolate milk
  Arms: 1% chocolate milk

SUMMARY:
The purpose of this experiment was to describe the effect of consuming 350 ml of 1% chocolate milk 60 minutes before a pizza meal on subjective appetite and short-term food intake when compared to cola, a fruit drink and a water control in normal weight and overweight/obese 9-14 year old boys and girls. It is hypothesized that 1% chocolate milk will increase meal time satiation to a greater extent than other sugars-sweetened commercially available beverages. Food intake will be measured 60 minutes after the consumption of 350 ml of water, fruit drink, cola or 1% chocolate milk.

ELIGIBILITY:
Inclusion Criteria:

* healthy boys and girls 9-14 years of age, stable weight, born at full term, normal birth weight

Exclusion Criteria:

* restricted diet, taking medications that affect food intake, significant learning, behavioral or emotional problems, food allergies to test treatments

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Food intake (kcal) | 60 min after the treatment

SECONDARY OUTCOMES:
Subjective appetite (in mm) | 0-90 min
  Subjective appetite by visual analogue scale (mm) measured at 0, 15, 30, 45, 60 and 90 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Applied Human Nutrition, Bedford, Nova Scotia, Canada